CLINICAL TRIAL: NCT06204692
Title: Computer Guided Versus Freehand Dental Implant Surgery: Randomized Controlled Clinical Trial
Brief Title: Computer Guided Versus Freehand Dental Implant Surgery
Acronym: dental implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Nermine Ramadan Mahmoud, Associated Professor, faculty of Dentistry, October 6 University, October 6 University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECO6U/29-2022; October6U (Other: October 6 University)
Record Dates: First submitted 2023-12-26; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Dental Implant
Keywords: virtual planning;; computer guided implants;; freehand implant;; dental implant
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Computer Guided Dental Implant Surgery. (Other): Computer Guided Dental Implant Surgery
  Interventions: Procedure: dental implant

INTERVENTIONS:
Procedure: dental implant — consisted of 6 patients where computer guided dental implant placement

SUMMARY:
This study's goal is to evaluate the efficacy of traditional rehabilitation with freehand implant implantation of partly or totally edentulous patients utilizing flapless or mini-flap procedures vs. 3D implant design software and specialized surgical templates.

DETAILED DESCRIPTION:
Patients with at least 7 mm of height and 4 mm of breadth in their bones, who needed at least two implants to be restored with a single prosthesis, were recruited one after the other. Patients were randomly assigned to two groups in a parallel group trial design. : Group I: consisted of 6 patients where computer guided dental implant placement and Group II: included six people who had dental implants placed manually. A temporary prosthesis was inserted into the implants right away, and four to six months later, a permanent prosthesis took its place.

Implant failures, marginal bone loss, number of therapy sessions, length of treatment, post-surgical pain and swelling, use of painkillers, surgical time, time needed to resolve problems, and patient satisfaction were among the outcome variables evaluated by a blinded, independent assessor. Patients were tracked for a full year.

ELIGIBILITY:
Inclusion Criteria:

* totally edentulous in one or both arches,
* with at least 7 mm of height and 4 mm of breadth in their bones as assessed by preoperative CBCT scans.
* patients between the ages of 35 and 65 who could give informed permission,
* Implants next to each other required to be positioned at least 3 mm apart from each other and 1.5 mm apart from the tooth.

Exclusion Criteria:

* Patients who have received radiation therapy to the head and neck region within the year prior to implantation,
* those who are receiving intravenous amino bisphosphonates,
* those who have untreated periodontitis,
* those with uncontrolled diabetes,
* pregnant women, or nursing mothers are among the general contraindications to implant surgery.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
marginal bone loss | 6 months postoperative
  Cone Beam Computed Tomography

SECONDARY OUTCOMES:
post-surgical pain and swelling | 7 days prior to implant placement
  Visual Analog Scale (10 represent maximum pain , 0 represent no pain)

CONTACTS AND LOCATIONS:
Locations (1):
- nermine Ramadan Mahmoud, Cairo, Egypt